CLINICAL TRIAL: NCT00303797
Title: A Phase I Study of the Raf Kinase/VEGFR Inhibitor BAY 43-9006 in Combination With the Proteasome Inhibitor PS-341 in Patients With Advanced Malignancies
Brief Title: Sorafenib and Bortezomib in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00124; MC0511; U01CA069912 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Stage III Multiple Myeloma; Stage IV Chronic Lymphocytic Leukemia; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — tanespimycin; Bortezomib; Sorafenib

ARMS (1):
- Treatment (bortezomib, sorafenib tosylate) (Experimental): GROUP I (solid tumors-dose-escalation group): Patients receive oral sorafenib twice daily on days 1-21 and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib and bortezomib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  GROUP II (multiple myeloma or chronic lymphocytic leukemia-maximum tolerated dose [MTD] group): Patients receive oral sorafenib at the MTD twice daily on days 3-21 of course 1 and on days 1-21 of each subsequent course. Patients also receive bortezomib IV over 3-5 seconds at the MTD on days 1, 4, 8, and 11.
  Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 17-N-allylamino-17-demethoxygeldanamycin/bortezomib; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: 17-N-allylamino-17-demethoxygeldanamycin/bortezomib
Drug: sorafenib tosylate
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
This phase I trial is studying the side effects and best dose of sorafenib and bortezomib in treating patients with advanced cancer. Sorafenib and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of cancer cells by blocking blood flow to the cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of sorafenib and bortezomib in patients with advanced malignancies.

II. To describe the toxicities associated with the combination of sorafenib and bortezomib.

III. To evaluate the therapeutic antitumor activity of the combination of sorafenib and bortezomib.

IV. To evaluate the effects of sorafenib on the disposition of bortezomib.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 groups according to disease type.

GROUP I (solid tumors-dose-escalation group): Patients receive oral sorafenib twice daily on days 1-21 and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib and bortezomib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

GROUP II (multiple myeloma or chronic lymphocytic leukemia-maximum tolerated dose [MTD] group): Patients receive oral sorafenib at the MTD twice daily on days 3-21 of course 1 and on days 1-21 of each subsequent course. Patients also receive bortezomib IV over 3-5 seconds at the MTD on days 1, 4, 8, and 11.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Cytologically or histologically proven unresectable solid tumor for which no curative treatment options exist (group I - dose-escalation phase)
  * Multiple myeloma or chronic lymphocytic leukemia requiring treatment (group II - maximum tolerated dose phase)

    * Failed ≥ 1 prior regimen
    * Non-secretory myeloma allowed
* No known standard therapy that is potentially curative or definitely capable of extending life expectancy exists
* Tumor amenable to serial sampling (group II)
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm^3 (75,000/mm^3 for patients with multiple myeloma [group II])
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (5 times ULN if liver involvement)
* Creatinine ≤ 1.5 times ULN (2.5 times ULN for patients with multiple myeloma [group II])
* Life expectancy ≥ 12 weeks
* No uncontrolled infection
* No New York Heart Association class III or IV heart disease
* No uncontrolled hypertension, labile hypertension, or history of poor compliance with antihypertensive medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No sensory peripheral neuropathy of any etiology > grade 1 or neuropathic pain of any etiology
* No active HIV infection requiring therapy
* No inability to swallow that would preclude use of oral medications
* No evidence of bleeding diathesis
* Medically capable and willing to provide biologic specimens as required (mandatory for patients in group II)
* Priorbortezomib allowed
* More than 3 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas) and recovered
* More than 4 weeks since prior immunotherapy or biologic therapy
* More than 2 weeks since prior steroid therapy (group II only)
* No prior anti-vascular endothelial growth factor therapy
* More than 4 weeks since prior full-field radiotherapy (2 weeks for limited-field radiotherapy)
* No prior radiation to > 25% of bone marrow
* More than 4 weeks since major surgery (e.g., laparotomy) (2 weeks for minor surgery)

  * Insertion of a vascular access device is not considered major or minor surgery
* No concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary other therapy considered investigational
* No concurrent prophylactic colony-stimulating factors
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial access devices allowed provided requirements for PT, INR, or PTT are met
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, and phenobarbital), rifampin, or Hypericum perforatum (St. John's Wort)
* No concurrent participation in any other study involving a pharmacologic agent (e.g., drugs, biologics, immunotherapy, or gene therapy), either for symptom control, or therapeutic intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
MTD as assessed by the number of patients with dose-limiting toxicity (DLT) using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | Observed for at least 3 weeks at a given dose level combination
  DLTs include: Hematologic: Grade 4 ANC for ≥5 days, Grade 4 anemia of any duration, or PLT <25,000 of any duration; Renal: Serum creatinine ≥2 times baseline or > 2x upper limit of normal if baseline levels normal; All other non-hematologic toxicities ≥grade 3 as per CTCAE v3.0 except fatigue; Any toxicities that caused dose delay of > 2 weeks of the intended next dose.
  MTD is the dose level below the lowest dose that induces DLT in at least one-third of patients (2 of 6 patients).
Toxicity as assessed by CTCAE v3.0 | Observed for at least 3 weeks at a given dose level combination
  Non-hematologic toxicities will be evaluated via the ordinal CTC standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via Common Toxicity Criteria standard grading.
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Antitumor activity as assessed by tumor measurement or evaluation of indicator lesion by computed tomography (CT) or magnetic resonance imaging (MRI) | Baseline, prior to each course (every 3 weeks) during dose escalation, every 6 weeks for solid tumors, and confirmatory scans at least 4 weeks following initial documentation of objective response
Effects of sorafenib on the disposition of bortezomib | From cohort II registration prior to each course
  Up to 20 patients with hematologic malignancies will be treated at the MTD to evaluate markers of drug activity and pharmacokinetics of this combination.

SECONDARY OUTCOMES:
Tumor response as assessed by CT or MRI using modified Response Evaluation Criteria in Solid Tumors (RECIST) | Baseline, every 3 weeks during dose escalation, every 6 weeks for solid tumors, and confirmatory scans at least 4 weeks following initial documentation of objective response
  CLL Modified RECIST:
  Measurable lesions: lesions that can be accurately measured in at least one dimension with longest diameter > 20 mm. With spiral CT scan, lesion must be > 10 mm in at least one dimension. Target lesions (up to 3) should be selected and a sum of the longest diameter (LD) for all will be the baseline sum LD. Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least 30% decrease in the sum of the longest diameter (LD) of target lesion taking as reference the baseline sum LD.
Best overall response as assessed using modified RECIST | Baseline until disease progression/recurrence
  CLL Progression (PD): As least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Duration of overall response | From the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date recurrent or progressive disease is documented
  Myeloma CR = Disappearance of M-protein from serum and urine, Bone marrow biopsy ≤5% plasma cells, No increase in lytic bone lesions, and Disappearance of soft tissue plasmacytomas. Patients who meet some, but not all, the criteria are classified as VGPR. Myeloma PR = 50-89% reduction of M-protein in serum and reduction of ≥90% or to <200 mg in 24-hour urinary light chain excretion (patients with non-secretory myeloma: a ≥50% reduction in plasma cells in a bone marrow aspirate), ≥50% reduction in soft tissue plasmacytoma, and No increase in number or size of lytic bone lesions.
Duration of stable disease | From the start of the treatment until the criteria for progression are met
  Myeloma PD: Increase of M-protein >25% above the lowest response level in serum or urine (absolute increase of at least 0.5 g/dL serum or 200 mg/24 hours urine); Patients with non-secretory myeloma: an increase in bone marrow plasmacytosis by 25% above the lowest remission value (absolute increase at least 10% bone marrow plasma cells); New soft tissue plasmacytomas or increase in size by 50% (and at least 1 cm); New lytic bone lesions or increase in the size of the existing bone lesions by 50% (and at least 1 cm); Development of hypercalcemia serum calcium >11.5 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kumar SK, Jett J, Marks R, Richardson R, Quevedo F, Moynihan T, Croghan G, Markovic SN, Bible KC, Qin R, Tan A, Molina J, Kaufmann SH, Erlichman C, Adjei AA. Phase 1 study of sorafenib in combination with bortezomib in patients with advanced malignancies. Invest New Drugs. 2013 Oct;31(5):1201-6. doi: 10.1007/s10637-013-0004-2. Epub 2013 Jul 26. PMID 23887852